CLINICAL TRIAL: NCT06772519
Title: Is It Possible to Reduce Surgical Pain and Nausea With Light Therapy? A Randomized Controlled, Non-Pharmacological Approach
Brief Title: Relieving Surgical Pain and Nausea With Light Therapy
Acronym: LITENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuran Ayşen Pamir Aksoy (Other)
Responsible Party: Sponsor-Investigator, Nuran Ayşen Pamir Aksoy, Assist. Prof., Acibadem University
Organization: Acibadem University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-18-687
Record Dates: First submitted 2025-01-10; First posted 2025-01-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Nausea and Vomiting, Postoperative
Keywords: colored-lens glasses; postoperative pain; organ donor; kidney transplantation; postoperative nausea; blue light; green light
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Group-Blue lens glasses (Experimental): Patients who assigned to this group will wear blue-lens glasses postoperatively (min 8 h in a day)
  Interventions: Device: blue colored lens glasses
- Study Group-Green lens glasses (Experimental): Patients who assigned to this group will wear green-lens glasses postoperatively (min 8 h in a day)
  Interventions: Device: green colored lens glasses
- Study Group-colorless (transparent) lens glasses (Placebo Comparator): Patients who assigned to this group will wear colerless (transparanet)-lens glasses postoperatively (min 8 h in a day)
  Interventions: Device: colorless (transparent) lens glasses
- Control group (No Intervention): Patients in this group will not be wearing any glasses. Patients will be asked to participate for postoperative pain and nausea assesment.

INTERVENTIONS:
Device: green colored lens glasses — Researchers will compare the blue-lens glasses and green-lens glasses groups to the transparent (colorless) glasses group and the non-glasses group to see if the colored lenses have an effect on postoperative pain and nausea.
  Other Names: green lens glasses
  Arms: Study Group-Green lens glasses
Device: blue colored lens glasses — Researchers will compare the blue-lens glasses and green-lens glasses groups to the transparent (colorless) glasses group and the non-glasses group to see if the colored lenses have an effect on postoperative pain and nausea.
  Other Names: blue lens glasses; colored lens glasses
  Arms: Study Group-Blue lens glasses
Device: colorless (transparent) lens glasses — Researchers will compare the blue-lens glasses and green-lens glasses groups to the transparent (colorless) glasses group and the non-glasses group to see if the colored lenses have an effect on postoperative pain and nausea.
  Arms: Study Group-colorless (transparent) lens glasses

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of colored (green and blue lens) glasses as a non-pharmacological method in relieving post-surgical pain and postoperative nausea in kidney donors. The main hypothesis it aims to test:

H1: Postoperative use of green-lensed glasses by patients who are kidney donors is effective in relieving surgical pain and postoperative nausea.

H2: Postoperative use of blue-lensed glasses by patients who are kidney donors is effective in relieving surgical pain and postoperative nausea.

Researchers will compare the blue-lens glasses and green-lens glasses groups to the transparent (colorless) glasses group and the non-glasses group to see if the colored lenses have an effect on postoperative pain and nausea.

Participants in the intervention groups will be asked

* to wear the glasses (according to their randomly assigned group (blue/green/colorless/), immediately after they admitted to the ward postoperatively, at least 8 hours in a day, until their discharge
* to respond the pain and nausea assessment (every 2 hours during postop day 1 and every 4 hours during postop day 2) until their discharge

Participants in the control group will be asked

- to respond the pain and nausea assessment (every 2 hours during postop day 1 and every 4 hours during postop day 2) until their discharge

DETAILED DESCRIPTION:
Since the hospital's architecture and clinical operation where the data will be collected have features that prevent patients from different groups from meeting, the single blind feature can be preserved. The pain assessment of the patients will be made with the numerical pain scale, and the nausea assessment will be made with the numerical nausea rating scale. In addition, data will be collected with the Patient Information Form prepared by the researchers in line with the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being a donor for kidney transplantation
* Not having an obstacle to wearing glasses
* Being able to communicate verbally

Exclusion Criteria:

* Being color blind • Developing post-operative complications during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | every 2 h during the post operative day1, and every 4 h during postoperative day 2.
  Post-operative pain level according to the numerical pain assessment scale
Post-operative nausea | every 2 h during the post operative day1, and every 4 h during postoperative day 2.
  Postoperative nausea level according to the numerical nausea rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Atakent Hospital, Istanbul, Atakent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided